CLINICAL TRIAL: NCT01553500
Title: Study of the Efficacy and Tolerability of Glucomannan on Children Affected by NAFLD
Brief Title: Glucomannan Effects on Children With Non-alcoholic Fatty Liver Disease
Acronym: GC-NASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Valerio Nobili, Principal Investigator, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPBG_GLUCO_2010
Record Dates: First submitted 2011-10-03; First posted 2012-03-14 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Metabolic Syndrome; Non Alcoholic Fatty Liver Disease; Insulin Resistance
Keywords: NAFLD; insulin resistance; children
MeSH Terms: conditions — Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Insulin Resistance | interventions — (1-6)-alpha-glucomannan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- glucomannan (Experimental)
  Interventions: Dietary Supplement: glucomannan
- placebo (Placebo Comparator)
  Interventions: Behavioral: lifestyle intervention

INTERVENTIONS:
Dietary Supplement: glucomannan — glucomannan is administered at dosage of 5g/day in form of biscuits (6 biscuits/day)
  Arms: glucomannan
Behavioral: lifestyle intervention — hypocaloric diet (25-30 Kcal/kg/day) or isocaloric (40-45 Kcal/kg/day) and physical activity
  Arms: placebo

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) has reached epidemic proportions and is rapidly becoming the one of most common causes of chronic liver disease in children. The pathogenesis of NAFLD is generally considered the result of a series of liver injuries, commonly referred as "multi-hit" hypothesis. Insulin resistance and increased serum levels of free fatty acids (FFAs) are considered the main primary hits that lead to the excessive lipid accumulation in hepatocytes resulting in steatosis.

Has been reported that a diet rich in high-viscosity fiber improves glycemic control and lipid profile, suggesting a therapeutic potential role in the treatment of NAFLD.

Aim of this study is to evaluate the efficacy and tolerability of glucomannan in children affected by non alcoholic fatty liver disease.

ELIGIBILITY:
Inclusion Criteria:

* informed consent by parents or legal tutor
* ALT levels <10 ULN
* hyperechogenicity at liver ultrasound examination suggestive of fatty liver
* INR < 1,3
* Albumin > 3 g/dl
* total bilirubin < 2,5 mg/dl
* no previous gastrointestinal bleeding
* no previous portosystemic encephalopathy
* normal renal function
* no HIV-HCV-HDV infection
* normal cell blood count

Exclusion Criteria:

* every clinical or psychiatric disease interfering with experimentation according to investigator's evaluation
* finding of active liver disease due to other causes
* corticosteroids, immunosuppressive drugs or chemotherapy in the 2 months before of the study
* alcohol consumption
* use of drugs known to induce steatosis or to affect body weight and carbohydrate metabolism
* finding of actual or previous level of alpha-fetoprotein > 50 ng/ml
* hepatocellular carcinoma
* diabetes mellitus type I

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in lipid profile | 6,12,18,24 months
  Evaluation of tryglicerides, total and LDL colesterol levels
Change from baseline in glycemic homeostasis | 6,12,18,24 months
  glycemic homeostesis will be evaluated through glycemia and insulinemia basal levels and after oral glucose tolerance test

SECONDARY OUTCOMES:
liver enzymes | 6,12,18,24 months
  evaluation of liver function test

CONTACTS AND LOCATIONS:
Overall Officials: Valerio Nobili, MD, Principal Investigator — Bambino Gesù Children's Hospital
Locations (1):
- Bambino Gesù Children's Hospital and Research Institute, Rome, Italy